CLINICAL TRIAL: NCT01839981
Title: A Pilot Study: Open-Label Clinical Trial of CPI-613 in Patients With Metastatic Pancreatic Adenocarcinoma and Poor Performance Status
Brief Title: CPI-613 in Treating Patients With Locally Advanced or Metastatic Pancreatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00023380; NCI-2013-00838 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CCCWFU 57113 (Other: Wake Forest University Health Sciences)
Record Dates: First submitted 2013-04-23; First posted 2013-04-25 (Estimated); Last update posted 2018-12-27 (Actual); Status verified 2018-06

CONDITIONS: Acinar Cell Adenocarcinoma of the Pancreas; Duct Cell Adenocarcinoma of the Pancreas; Recurrent Pancreatic Cancer; Stage III Pancreatic Cancer; Stage IV Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — devimistat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (6,8-bis(benzylthio)octanoic acid) (Experimental): Patients receive 6,8-bis(benzylthio)octanoic acid IV over 2 hours on days 1-5 of week 1 (pre-course 1 only), days 1 and 4 of weeks 2 and 3 (course 1 only), and days 1 and 4 of weeks 1-3 (courses 2-6). Treatment repeats every 4 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: 6,8-bis(benzylthio)octanoic acid

INTERVENTIONS:
Drug: 6,8-bis(benzylthio)octanoic acid — Given IV
  Other Names: alpha-lipoic acid analogue CPI-613; CPI-613

SUMMARY:
This pilot clinical trial studies 6,8-bis(benzylthio)octanoic acid in treating patients with locally advanced or metastatic pancreatic cancer. Drugs used in chemotherapy, such as 6,8-bis(benzylthio)octanoic acid, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine initial estimates of overall survival (OS).

SECONDARY OBJECTIVES:

I. To determine response rate. II. To determine progression free survival (PFS).

OUTLINE:

Patients receive 6,8-bis(benzylthio)octanoic acid intravenously (IV) over 2 hours on days 1-5 of week 1 (pre-course 1 only), days 1 and 4 of weeks 2 and 3 (course 1 only), and days 1 and 4 of weeks 1-3 (courses 2-6). Treatment repeats every 4 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Histologically and cytologically proven locally advanced or metastatic pancreatic adenocarcinoma that is not amenable to surgery, radiation, or combined modality therapy with curative intent, and has failed or is not eligible for available chemotherapies
* Local, locally-advanced, or metastatic disease documented as having shown progression on a scan (e.g., computed tomography [CT], magnetic resonance imaging [MRI])
* Measurable tumor according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria with at least one unidimensionally measurable target lesion
* No evidence of biliary duct obstruction, unless obstruction is controlled by local treatment or, in whom the biliary tree can be decompressed by endoscopic or percutaneous stenting with subsequent reduction in bilirubin to below 1.5 x upper level of normal (ULN)
* No acute toxic effects from previous treatment superior to grade 1 at the start of the study
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-3
* Expected survival > 3 months
* Women of child-bearing potential (i.e., women who are pre-menopausal or not surgically sterile) must use accepted contraceptive methods (abstinence, intrauterine device [IUD], oral contraceptive or double barrier device) during the study, and must have a negative serum or urine pregnancy test within one week prior to treatment initiation
* Fertile men must practice effective contraceptive methods during the study, unless documentation of infertility exists
* Granulocyte count >= 1500/mm^3
* White blood cell (WBC) >= 3500 cells/mm^3 or >= 3.5 bil/L
* Platelet count >= 100,000 cells/mm^3 or >= 100 bil/L
* Absolute neutrophil count (ANC) >= 1500 cells/mm^3 or >= 1.5 bil/L
* Hemoglobin >= 9 g/dL or >= 90 g/L
* Aspartate aminotransferase (AST)/(serum glutamic oxaloacetic transaminase [SGOT]) =< 3 x upper normal limit (UNL), alanine aminotransferase (ALT)/(serum glutamate pyruvate transaminase [SGPT]) =< 3 x UNL (=< 5x UNL if liver metastases present)
* Bilirubin =< 1.5 x UNL
* Serum creatinine =< 2.0 mg/dL or 177 umol/L
* International normalized ratio (INR) must be =< 1.5
* No evidence of active infection and no serious infection within the past month
* Mentally competent, ability to understand and willingness to sign the informed consent form

Exclusion Criteria:

* Patients receiving any other standard or investigational treatment for their cancer, or any other investigational agent for any indication within the past two weeks prior to initiation of CPI-613 (6,8-bis(benzylthio)octanoic acid) treatment
* Serious medical illness that would potentially increase patients' risk for toxicity
* Any active uncontrolled bleeding and any patients with a bleeding diathesis (e.g., active peptic ulcer disease)
* Pregnant women, or women of child-bearing potential not using reliable means of contraception
* Lactating females
* Fertile men unwilling to practice contraceptive methods during the study period
* Life expectancy less than 3 months
* Any condition or abnormality which may, in the opinion of the investigator, compromise the safety of patients
* Unwilling or unable to follow protocol requirements
* Dyspnea with moderate exertion
* Patients with pleural or pericardial effusions
* Active heart disease including but not limited to symptomatic congestive heart failure, symptomatic coronary artery disease, symptomatic angina pectoris, symptomatic myocardial infarction, also patients with a history of myocardial infarction that is < 1 year prior to registration, or patients with previous congestive heart failure (< 1 year prior to registration) requiring pharmacologic support or with left ventricular ejection fraction < 45%
* A history of additional risk factors for torsade de pointes (e.g., heart failure, hypokalemia, family history of long QT syndrome)
* Evidence of active infection, or serious infection within the past month
* Patients with known human immunodeficiency virus (HIV) infection
* Patients who have received cancer immunotherapy of any type within the past 2 weeks prior to initiation of CPI-613 treatment
* Requirement for immediate palliative treatment of any kind including surgery
* Patients that have received a chemotherapy regimen with stem cell support in the previous 6 months
* Prior illicit drug addiction
* Any condition or abnormality which may, in the opinion of the investigator, compromise the safety of the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-07; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Overall Survival | From the first dose of 6,8-bis(benzylthio)octanoic acid to death, assessed up to 3 years
  Survival curves for OS will be estimated using Kaplan-Meier techniques.

SECONDARY OUTCOMES:
Response rate | Up to 3 years
  The proportion of patients who are complete response (CR), partial response (PR), stable disease (SD), or progressive disease (PD) will be presented. The proportion of responders will be estimated as the percent of patients who are CR or PR. A 95% confidence interval will be included.
Progression Free Survival | From the first dose of 6,8-bis(benzylthio)octanoic acid to disease progression (DP) or death due to any cause, assessed up to 3 years
  Survival curves for PFS will be estimated using Kaplan-Meier techniques.
Safety profile assessed using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 | Up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Caio Rocha Lima, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Comprehensive Cancer Center of Wake Forest University, Winston-Salem, North Carolina, United States